CLINICAL TRIAL: NCT01178619
Title: Sonographic Differences in Brain Measurements Between Normal and Intrauterine Growth Restriction (IUGR) Fetuses
Status: Withdrawn | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10095-2010CTIL
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Intra-uterine Growth Restriction
Keywords: IUGR fetuses; symmetrical IUGR; asymmetrical IUGR

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (3):
- AGA
- symmetrical IUGR
- asymmetrical IUGR

SUMMARY:
Intrauterine growth restriction is being suspected in cases where the fetal estimated weight is less then the 10 th percentile for its gestational age. Abdominal circumference is the most influenced measurement in this cases. Head circumference on the other hand can be or not be influenced. Previous studies have shown that transverse cerebellar diameter (TCD) is constant to gestational age and is not influenced by IUGR.Other showed lower TCD in IUGR fetuses. We would like to study the differences in cerebellar, vermian and corpus callosum growth between normal to IUGR fetuses and between symmetrical and asymmetrical IUGR. In this observational study we will include pregnant women between 28-37 gestational week with a singleton otherwise normal pregnancies. We will measure the fetal TCD, vermian distances and the CC, abdominal circumference, head circumference and femur length. we will compeer these measurements according to the following groups:normal fetuses, symmetrical and asymmetrical IUGR.

ELIGIBILITY:
Inclusion Criteria:

* singleton,
* 28-37 GA,
* well dated pregnancy.

Exclusion Criteria:

* multifetal pregnancies,
* no first trimester dating,
* fetuses with known chromosomal or structural anomalies.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pregnant women 28-37 GA, singleton, otherwise normal fetuses
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Actual)